CLINICAL TRIAL: NCT07043803
Title: Reduction of Anticholinergic Medications Project (RAMP) Among Persons With Schizophrenia or Other Psychiatric Disorders Across UPMC Behavioral Healthcare Partner Organizations Using a Stepped-wedge, Randomized Trial Study Design.
Brief Title: Reduction of Anticholinergic Medications Among Persons With Schizophrenia or Other Psychiatric Disorders
Acronym: RAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STUDY24120064; UL1TR001857 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Schizophenia Disorder; Schizoaffective Disorder; Bipolar Disorder; Psychiatric Disorders
Keywords: schizophrenia; implementation study; serious mental illness; psychiatric disorders; anticholinergic medication deprescription; anticholinergic side effects; Quality of life
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Mental Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The investigators will use a stepped-wedge open-cohort single arm trial design, where each of the four sites is randomized 2 to 6 weeks apart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anticholinergic Medication Reduction (Other)
  Interventions: Other: Reduction of anticholinergic medication

INTERVENTIONS:
Other: Reduction of anticholinergic medication — Shared decision making between the patient and prescriber will determine the timing and speed of reduction over a period of 12 to 16 weeks. Some patients will be discontinued from these anticholinergic medications (benztropine/trihexyphenidyl), others will be tapered from their original dosage but not completely discontinued, and some patients may not be able to taper the anticholinergic medications at all.

SUMMARY:
The goal of this study is to reduce Anticholinergic Medication (ACM) in persons with psychoses or serious mental illness, when these medications are no longer needed.

DETAILED DESCRIPTION:
Based on the investigator's preliminary work, the investigators will utilize a combination of administrative, prescriber and patient buy-in to reduce Anticholinergic Medication (ACM), when these medications are no longer needed, as evidence-based practice. Previously developed materials and tools from the investigator's earlier work include an ACM side-effect scale (the Pittsburgh Anticholinergic Symptoms Scale, PASS v2.0), a patient-facing information leaflet reviewing the risks of long-term ACM use, and a Clinical Guide for deprescribing. These, as well as education on the Anticholinergic Medication Burden (ACMB) reduction protocol will be provided to prescribers at initiation of each site. The clinical pharmacist on the team will train staff at each site to compute and record the Anticholinergic Cognitive Burden and use the PASS to assess ACM side effects. The investigators will train the staff members to administer the Memory Impairment Screen, a verbal working memory task.

The Principal Investigator (PI) and members of the study team will work with the healthcare teams at each site using case examples of 'how to reduce and/or stop anticholinergic medications" and maintain office hours on a scheduled basis to problem-solve, trouble-shoot and/or manage the medication reduction process and clinical issues that emerge. The PI and members of the study team will train the healthcare teams at each site to examine eligible patients for extra pyramidal symptoms and in the use of a shared decision-making approach in this effort to reduce anticholinergic medications.

Based on considerable interest from our healthcare partners, and in the absence of any randomized studies, the investigators intend to use a stepped-wedge, randomized trial study design to implement this protocol for eligible patients in each of the participating clinics. In addition to affirming earlier positive clinical outcomes in the preliminary work, the investigators intend to assess barriers to and facilitators of anticholinergic medication burden reduction implementation to inform the emerging evidence-based practice.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 years or older
2. have a chart DSM V diagnosis of schizophrenia spectrum or schizoaffective or bipolar disorder or any other mental illness disorder
3. have received ACM and antipsychotic medications for 6 months or more
4. are considered to be clinically stable (by the patient's healthcare team) for 3 months or more
5. the ACM (e.g. benztropine and/or trihexyphenidyl) is being used to treat EPS associated with antipsychotic medications.
6. on an examination using the modified Simpson-Angus Extrapyramidal Symptoms Scale (head dropping and leg pendulousness items are dropped), no single item rated at 3 or 4.
7. able and willing to sign the approved informed consent document.

Exclusion Criteria:

1. patients with ongoing Parkinsonian symptoms who require ACM meds for countering EPS side effects based on the Simpson-Angus Scale score cutoffs.
2. if the clinicians treating the potentially eligible patients consider them to be clinically unstable or if drug-addiction is the focus of treatment and participation in ACM de-prescription protocols is considered risky, the team will defer to the treating clinicians to exclude participants.
3. The same exclusions will apply to those persons undergoing medical procedures and treatments that make participation in this ACM deprescription trial unwise per the treating team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of Anticholinergic Medications | From enrollment to final visit. The final visit can vary for each participant and can be up to 16 weeks following the first baseline visit.
  For the primary outcome, reduction of anticholinergic medications (benztropine and/or trihexyphenidyl) will be computed as a percentage reduction from baseline. Those participants who discontinued fully will be considered as having a 100% reduction, and those who tapered but did not discontinue will be computed as a percentage reduction from baseline, and those participants who did not discontinue at all will be considered to have a zero-percentage reduction. This anticholinergic medication reduction will be computed at the end of the study for each participant and summed for all study participants.

SECONDARY OUTCOMES:
Auditory Verbal Learning and Recall | Enrollment to final visit. This can vary for each participant after Visit 1 (baseline) and be up to 16 weeks.
  The Memory Impairment Screen (MIS) is being used to assess auditory verbal learning and free or cued recall memory. Lower scores are indicative of poorer learning and memory; the total scores range from 0 to 8. Scores of 5 through 8 generally indicate no memory impairment, scores of 4 or lower indicate memory concerns.
The Pittsburgh Anticholinergic Symptoms Scale v2.0 (PASS) | Enrollment to final visit which can vary for each participant after Visit 1 (baseline) and can be up to 16 weeks.
  This is a self-report scale guided by clinicians for participants to fill out regarding the occurrence of side effects which may be associated with anticholinergic medications like benztropine and/or trihexyphenidyl. These include symptoms such as dry mouth, blurred vision, difficulty urinating, constipation, fast heartbeat or confusion/memory problems. Each item is anchored to the last week for recall by the patient and is rated from 0 (no side effects) to 6 (all the time and every day). The total score is computed by adding the 6 items, and ranges from a score of zero (none) to 36 (maximum), higher scores indicate worse anticholinergic effects. The last two items, intensity (overall severity, considering the six individual items), and impact on day-to-day functioning, are also scored 0 (none) to 6, 6 being intolerable or unable to function. The last two items are computed separately from the top 6 individual items and range from 0 (none) to 12 (severe or intolerable).
Anticholinergic Cognitive Burden Scale (ACB) | Enrollment to final visit which can vary for each participant after Visit 1 (baseline) and can be up to 16 weeks.
  This widely used scale provides a score of the anticholinergic medication burden in an individual participant, and the potential impact on cognition in an individual patient. The scale was developed by expert consensus and is based on clinical evidence of an individual anticholinergic medication's impact on cognition either from the literature, or in vivo or in vitro data, or available data from the manufacturer, and/or the ability to induce delirium. Each medication is scored from a minimum of 1 to a maximum of 3, with 3 indicating highly anticholinergic medications (e.g. benztropine or trihexyphenidyl). The scale authors have suggested a score of 3 or greater is clinically significant for anticholinergic impact on cognition. For purposes of this clinical study, in addition to the original list of anticholinergic medications, the investigators have added an updated medication list (following market approval of psychotropic drugs) to the original list with anticholinergic properties.

CONTACTS AND LOCATIONS:
Overall Officials: Professor of Psychiatry, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Western Behavioral Health of the Alleghenies, Altoona, Pennsylvania
  - UPMC Western Behavioral Health at Safe Harbor, Erie, Pennsylvania
  - Western Behavioral Health Mon Yough, McKeesport, Pennsylvania
  - Comprehensive Recovery Services (Pittsburgh) of Western Psychiatric Hospital, Ambulatory Clinics and Residential Programs - UPMC, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lupu AM, MacCamy KL, Gannon JM, Brar JS, Chengappa KNR. Less is more: Deprescribing anticholinergic medications in persons with severe mental illness. Ann Clin Psychiatry. 2021 May;33(2):80-92. doi: 10.12788/acp.0019. Epub 2021 Feb 1. PMID 33878282
- [Background] Lupu AM, Clinebell K, Gannon JM, Ellison JC, Chengappa KNR. Reducing Anticholinergic Medication Burden in Patients With Psychotic or Bipolar Disorders. J Clin Psychiatry. 2017 Nov/Dec;78(9):e1270-e1275. doi: 10.4088/JCP.16m11269. PMID 29178683